CLINICAL TRIAL: NCT00419874
Title: Blood- Brain Barrier Permeability in Neurological Patients: Anatomical, Neurophysiological, and Clinical Characteristics
Brief Title: Characteristics of Blood- Brain Barrier Permeability in Neurological Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Other Study IDs: SOR444206CTIL
Record Dates: First submitted 2007-01-07; First posted 2007-01-09 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2006-11

CONDITIONS: Traumatic Brain Injury; Cerebral Infarction; Cerebral Hemorrhage
Keywords: Blood-brain barrier; Post traumatic epilepsy; Seizures
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Infarction; Cerebral Hemorrhage; Epilepsy, Post-Traumatic; Seizures

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The main goal of the present study is to challenge the hypothesis that blood- brain barrier disruption following brain injury increases the risk for long-term disability, development of brain dysfunction, epileptic seizures and neuroanatomical alterations.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is one of the most common traumatic events, occurring in approximately 200 per 100,000, and is a known risk factor for later development of epileptic seizures. This occurs in up to 17% of TBI patients, and accounts for approximately 20% of symptomatic epilepsies (Annegers, JF. et al, 1998). Typically, post-traumatic epilepsy (PTE) develops or several weeks but even years after the event. PTE is often chronic and poorly controlled pharmacologically. Although several factors have been attributed to an increased risk of developing PTE (e.g. severity of trauma, type of brain injury, time to the appearance of first seizure), the mechanisms underlying it remain unknown. Similar to TBI, ischemic injuries, most frequently occurring in the elderly population are the main cause of new onset epilepsy in this age group. It is still not known what are the risk factors and mechanisms underlying post-ischemic epilepsy.

Under normal conditions the central nervous system is protected by the operation of the blood- brain barrier (BBB). Following brain injury (either traumatic or ischemic) the BBB is known to disrupt, leading to focal edema and altered extracellular composition. We have recently established methods for quantitative evaluation of the integrity of the BBB using magnetic resonance imaging (MRI) brain scans. Using these methods we are able to identify BBB disruption in patients suffering from various pathologies (Tomkins, O. et al. 2001; Avivi, E. et al. 2004). Such altered permeability may last up to years following the acute event and was found to correlate to areas of abnormal neurological function (Korn, A. et al. 2005)

In recent work using an animal model, we have shown that following focal disruption of the BBB a focus of epileptiform activity is generated within several days. Such pathological activity remains for several weeks, long after the BBB has retained its former function (Seiffert, E. et al. 2004; Iven, S. et al. 2006). Furthermore, this condition may later lead to anatomical alterations as seen by brain MRI scans, as well as in histological sections. Such animals further suffer from functional deterioration and neuronal degeneration in the disrupted region (Tomkins, O. et al. 2006).

In this work we will test the hypothesis that BBB disruption following brain injury increases the risk for long-term disability, development of brain dysfunction, epileptic seizures and neuroanatomical alterations. For that we will combine a prospective and retrospective study in patients following cerebral cortical injury (traumatic, hemorrhagic or ischemic). Clinical, functional and anatomical measures will be obtained in addition to BBB permeability measures.

ELIGIBILITY:
Inclusion Criteria:

* One week following:

  * Traumatic Brain Injury
  * Cerebro- Vascular Accident
* Subsequent brain CT showed cerebral cortex injury.

Exclusion Criteria:

* A known ailment of the central nervous system.
* Use of medications or illicit drugs that significantly affect the central nervous system.
* tourist or temporary residents not available for follow-up.
* For MRI examinations: heart pacemaker, metal implants, or metal shrapnel.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Overall Officials: Alon Friedman, MD/PhD, Principal Investigator — Soroka University Medical Center; Ilan Shelef, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Background] Tomkins O, Friedman O, Ivens S, Reiffurth C, Major S, Dreier JP, Heinemann U, Friedman A. Blood-brain barrier disruption results in delayed functional and structural alterations in the rat neocortex. Neurobiol Dis. 2007 Feb;25(2):367-77. doi: 10.1016/j.nbd.2006.10.006. Epub 2006 Dec 22. PMID 17188501
- [Background] Ivens S, Kaufer D, Flores LP, Bechmann I, Zumsteg D, Tomkins O, Seiffert E, Heinemann U, Friedman A. TGF-beta receptor-mediated albumin uptake into astrocytes is involved in neocortical epileptogenesis. Brain. 2007 Feb;130(Pt 2):535-47. doi: 10.1093/brain/awl317. Epub 2006 Nov 21. PMID 17121744
- [Background] Dreier JP, Jurkat-Rott K, Petzold GC, Tomkins O, Klingebiel R, Kopp UA, Lehmann-Horn F, Friedman A, Dichgans M. Opening of the blood-brain barrier preceding cortical edema in a severe attack of FHM type II. Neurology. 2005 Jun 28;64(12):2145-7. doi: 10.1212/01.WNL.0000176298.63840.99. PMID 15985592
- [Background] Seiffert E, Dreier JP, Ivens S, Bechmann I, Tomkins O, Heinemann U, Friedman A. Lasting blood-brain barrier disruption induces epileptic focus in the rat somatosensory cortex. J Neurosci. 2004 Sep 8;24(36):7829-36. doi: 10.1523/JNEUROSCI.1751-04.2004. PMID 15356194